CLINICAL TRIAL: NCT06507865
Title: Characterization of Mid-term Post Market Clinical Follow Up of GORE® TAG® Thoracic Branch Endoprosthesis Facilitated Aortic Arch and Descending Aorta Intervention
Brief Title: Post Market Registry for GORE® TAG® Thoracic Branch Endoprosthesis
Status: Recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: TGR 23-02TB
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Aneurysm; Dissection, Aortic; TAA Thoracoabdominal Aortic Aneurysm; Thoracic Aortic Aneurysm; Transection Aorta
Keywords: TEVAR; Aneurysm; Dissection; Aorta; Endovascular stent graft; Thoracic branch endoprosthesis
MeSH Terms: conditions — Aneurysm; Aortic Dissection; Aortic Aneurysm, Thoracoabdominal; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- GORE® TAG® Thoracic Branch Endoprosthesis: Patients treated with the TBE Device
  Interventions: Device: GORE® TAG® Thoracic Branch Endoprosthesis

INTERVENTIONS:
Device: GORE® TAG® Thoracic Branch Endoprosthesis — Patients presenting with thoracic vascular disease that may benefit from the placement of TBE device. The target registry population is patients who are treated with TBE at participating sites. TBE treatment is qualified as receiving the TBE aortic component, at a minimum.
  Other Names: TBE device

SUMMARY:
The goal of this observational study is to collect mid-term post-market clinical follow-up data of GORE® TAG® Thoracic Branch Endoprosthesis used according to the standard medical practice in patients presenting with vascular disease. This registry aims to answer questions related to the efficacy and safety of GORE® TAG® Thoracic Branch Endoprosthesis.

DETAILED DESCRIPTION:
The purpose of the GORE® TAG® Thoracic Branch Endoprosthesis Registry is to collect real-world data for this device. Due to the nature of the registry, patient selection, diagnostic imaging, and treatment interventions will be determined by physicians based on standard clinical practice. Therefore, the Sponsor will not be outlining requirements that would influence healthcare decisions.

Participants will be asked to return for regular scheduled visits as requested by their surgeon. Patients will report any issues they may have regarding the device or surgery to their surgeon/doctor.

ELIGIBILITY:
Inclusion Criteria:

Patient or legally authorized representative (LAR) provides written authorization and/or consent per institution and geographical requirements Patient has been or is intended to be treated with an eligible registry device Patient is age ≥ 18 years at time of informed consent signature.

Exclusion Criteria:

Patient who is, at the time of consent, unlikely to be available for standard of care (SOC) follow-up visits as defined by the site's guidelines and procedures.

Patient with exclusion criteria required by local law. Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study within 12 months of Together Registry enrollment. Subjects cannot be enrolled in another Together Registry module protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Registry participants are derived from patients presenting with vascular disease that may benefit from the placement of an endovascular stent graft. The target registry population is patients who are treated with TBE at participating sites. Only patients who meet all the inclusion and none of the exclusion criteria will be included in the registry.
  The registry has been designed with broad eligibility criteria to optimize the visibility of overall registry device use. An integral requirement to the target subject population is that the decision to use a TBE product has been made prior to considering the patient for possible registry participation. The TBE registry population will be defined as a successful recipient of TBE at the end of the index procedure.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Deployment Technical Success | Time of Surgery
  Successful access, delivery, and accurate deployment of the device to the intended location, and retrieval of the delivery system. The absence of any additional corrective procedure related to the device, procedure, or withdrawal of the delivery system. Events will not include interventions at the access site(s), lumbar drains to address spinal cord ischemia, or additional interventions to address non-treatment areas.
Lesion-related Mortality | Day 30 through Year 2
  Death related to the index endovascular procedure or following conversion to open repair and death related to a complication from a secondary procedure associated with the index lesion or registry device.
  Any death where the treated disease / index lesion or registry device caused or significantly contributed to the death, including lesion-rupture, aortic-related complications, disease progression involving the index lesion.
Lesion Rupture (treated area) | Time of Surgery through Year 2
  Rupture in the treated segment of the vessel (e.g., aorta or branch) verified with direct observation or CT / CTA scan.
Lesion Enlargement (treated area) | Time of Surgery through Year 2
  An increase in maximum vessel (e.g., aorta or treated branch) diameter of > 5 mm in the region encompassed by the initial lesion as compared to baseline using orthogonal (i.e., perpendicular to the centerline) measurements on CT / CTA scans.
Endoleaks (Type I-V) | Time of Surgery through Year 2
  Perfusion of a treated lesion identified through imaging analysis.
Device Migration | Time of Surgery through Year 2
  Longitudinal movement of all or part of the device for a distance ≥ 10 mm, as confirmed by CTA scan, relative to anatomical landmarks and device positioning at the first post-operative CTA scan.
Loss of Aortic / Branch Patency | Time of Surgery through Year 2
  No flow or contrast detected through the implanted aortic and/or branch component (for branched devices) confirmed with imaging and/or direct observation.
Stroke | Time of Surgery through Year 2
  Stroke is the acute onset of symptoms consistent with focal or multifocal central nervous system (CNS) injury caused by vascular blockage resulting in ischemia or vascular rupture resulting in hemorrhage, that either persists for > 24 hours or until death or symptoms lasting < 24 hours, with pathology or neuroimaging confirmation of CNS infarction.
Paraplegia | Time of surgery through Day 30
  New onset spinal cord injury rendering a subject non-ambulatory.
Paraparesis | Time of surgery through Day 30
  New onset spinal cord injury causing a minor motor deficit of the lower extremities.
New Onset Renal Failure | Time of surgery through Day 30
  New onset sustained renal failure identified within 30 days of the index endovascular procedure, combined with requiring dialysis for > 4 weeks.
Renal Function Deterioration | Time of surgery through Year 2
  New onset of a decrease in eGFR > 30% following treatment when compared to baseline eGFR.
Device Integrity Events | Time of Surgery through Year 2
  wire fractures, stent kinking, disruption/tears in the graft component, or stent compression or invagination identified through imaging analysis.
Reintervention | Time of Surgery through Year 2
  Additional surgical or interventional procedure related to the treated disease / index lesion, the registry device, or to the treatment / procedure.
  This may include surgical or interventional treatment for endoleaks, access site(s) complications, disease progression (including interventions to address issues related to non-treated area of the index lesion, such as bare stent implantation to address bowel ischemia associated with aortic dissection), spinal drains for Spinal Cord Injury (SCI) management, or conversion to open surgery.

SECONDARY OUTCOMES:
Access-related Complications | Time of Surgery through Year 2
  Complications associated with the access sites used during treatment and any subsequent unplanned access-related reinterventions. This may include pseudoaneurysm, hematoma, thrombosis, or complications associated with percutaneous closure devices.
Transient Ischemic Attack (TIA) | Time of Surgery through Year 2
  Transient focal neurological signs or symptoms (lasting <24 h) presumed to be due to focal brain ischemia but without evidence of acute infarction by neuroimaging or pathology (or in the absence of imaging)
Life Threatening Bleed | Time of Surgery through Year 2
  An event leading to either diagnosed hypovolemic shock, required four or more packed red blood cell units or directly led to subject death.
Upper Extremity Ischemia | Time of Surgery through Year 2
  Clinically-reported, device-related ischemia not evident at the time of the index procedure with CTA-verified branch vessel compromise (i.e., malperfusion)
False Lumen Status - Treated Segment | Time of Surgery through Year 2
  Status of the false lumen within the segment of the aorta initially treated with an endovascular stent graft. It is divided in patent, partial thrombosis and complete thrombosis.
False Lumen Status - Untreated Segment | Time of Surgery through Year 2
  Status of the false lumen outside of the segment of the aorta initially treated with an endovascular stent graft. It is divided in patent, partial thrombosis and complete thrombosis.
False Lumen Perfusion | Time of Surgery through Year 2
  Flow into the false lumen via Type IA entry flow, Type IB entry flow, Type II entry flow and Type R entry flow.

CONTACTS AND LOCATIONS:
Locations (20):
- Medizinische Universität Wien, Vienna, Austria
- Rigshospitalet University Hospital, Copenhagen, Denmark
- Germany (4):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - University of Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Münster, Münster
- Greece (2):
  - Evangelismos General Hospital, Athens
  - Laiko General hospital of Athens, Athens
- Italy (5):
  - Policlinico di Sant'Orsola, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - IRCCS Ospedale Policlinico San Martino, Genova
  - AOU Padova, Padua
  - Azienda Ospedaliera "G. Brotzu", Selargius
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - Radboud UMC, Nijmegen
- Spain (2):
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Hospital Universitario Miguel Servet, Zaragoza
- Skane University Hospital, Malmo, Sweden
- United Kingdom (2):
  - St Thomas' Hospital, London
  - St Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared will be pseudo-anonymized with subject names and birthdates removed.
Time Frame: Sharing of IPD will not routinely be performed and is contingent on an assessment of the researcher's proposal for novelty or value in advancing educational, quality or medical practice objectives in use of this data.
Access Criteria: See above